CLINICAL TRIAL: NCT02515474
Title: A Long Term Comparison of Laparoscopic Common Bile Duct Exploration and Cholecystectomy Versus Sequential ERCP Followed by Cholecystectomy for Choledocholithiasis: a Multicenter Prospected Non-randomized Controlled Study
Brief Title: Comparison of LCBDE vs ERCP + LC for Choledocholithiasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hepatopancreatobiliary Surgery Institute of Gansu Province (Other)
Responsible Party: Principal Investigator, Xun Li, professor of surgery, Hepatopancreatobiliary Surgery Institute of Gansu Province
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Complications of LCBED vs ERCP
Record Dates: First submitted 2015-07-30; First posted 2015-08-04 (Estimated); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Choledocholithiasis
Keywords: Cholangiopancreatography; Endoscopic; Common bile duct; Complication; Recurrence; Laparoscopic
MeSH Terms: conditions — Choledocholithiasis; Recurrence | interventions — Laparoscopy; Endoscopy; Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LCBDE group (single step) (Active Comparator): Choledocholithiasis patient, after Laparoscopic Cholecystectomy (LC) to remove the gallbladder, Laparoscopic Common Bile Duct Exploration (LCBDE) was performed for removing the bile duct stone(s) in laparoscopy. Choledochoscope detection or cholangiograms should be chosen as a method of obtain stone clearance. T-tube was acceptable if needed.
  Interventions: Procedure: Laparoscopy
- ERCP group (sequential step) (Active Comparator): Choledocholithiasis patient, Endoscopic Retrograde cholangiopancreatography (ERCP) was performed for removing the bile duct stone(s) in endoscopy prior to Laparoscopic Cholecystectomy (LC). Sphincterotomy (EST) and Endoscopic papillary balloon dilatation (EPBD) can be chosen accordingly. The laparoscopic cholecystectomy was subsequently performed as soon as technically feasible following the ERCP in one month.
  Interventions: Procedure: Endoscopy

INTERVENTIONS:
Procedure: Laparoscopy — After removing the gallbladder, Laparoscopic common bile duct exploration (LCBDE) was performed by one fulltime attending in laparoscopy in a routine fashion. Access from the opening of the anterior wall of common bile duct or from the dilated cystic duct was acceptable, removed stone(s) and irrigated the duct followed by choledochoscope detection simultaneously. Cholangiograms were also can be a alternative method to obtain stone clearance. If needed, all fluoroscopy was performed by the principal author in the presence of and concurrence with the ERCP endoscopist. Once the LCBDE was completed, the incision of the bile duct was sewed intermittently by absorbed threads, or ligated cystic duct. T-tube was acceptable if needed.
  Other Names: Laparoscopic common bile duct exploration (LCBDE)
  Arms: LCBDE group (single step)
Procedure: Endoscopy — Initially endoscopic retrograde cholangiopancreatography (ERCP) was performed by a fulltime attending and concurrence of the principal author in endoscopy. Patients randomized to ERCP+ LC group were scheduled to undergo the endoscopic procedure using fluoroscopy in the endoscopy center under moderate sedation (principally intravenous midazolam and meperidine) prior to the intended laparoscopy. Gastric intestinal atony during ERCP was routinely achieved using scopolamine butylbromide injection. Sphincterotomy (EST) and Endoscopic papillary balloon dilatation (EPBD) can be choose accordingly. The laparoscopic cholecystectomy was subsequently performed as soon as technically feasible following the ERCP in one month.
  Other Names: Endoscopic Retrograde cholangiopancreatography (ERCP)
  Arms: ERCP group (sequential step)

SUMMARY:
Protection of Oddi's sphincter remains a huge argument especially in the long term complications like common bile duct stone recurrence or cholangitis after ERCP, which determined to destroy the sphincter of Oddi. The purpose of this study is to compare the long-term outcomes of ERCP sequential LC versus LCBDE for choledocholithiasis.

DETAILED DESCRIPTION:
Cholelithiasis, a common etiology factor responsible for abdominal pain, is highly prevalent worldwide. According to data from general investigation, the morbidity of cholelithiasis differs from 2.36% to 42% in different areas, and about 5% to 29% (average 18%) of all cholelithiasis cases have both gallbladder stone and common bile duct stone. In the population with age above 70 years old, 30% of which suffers from gallbladder stone in China. A causal link between the development of gallbladder stone and common bile duct stone is that 10% to 15% of gallstone patients have high potential to develop secondary common bile duct stone. In 1987, the laparoscopic cholecystectomy (LC) came into being as a revolutionary surgical method. With minimally invasive effect and high safety, LC was soon accepted as a 'Golden standard' for the treatment of gallbladder stone. Endoscopic sphincterotomy (EST) was firstly reported by Kawai and Classen in 1970. As of now, the combination of EST with other endoscopic techniques, such as basket extraction, balloon dilation and lithotripsy, have significantly improved the stone removal rate from 85% up to 90%, and ERCP has been considered as the optimal method in regard to CBD stone treatment. In 1991, the laparoscopic common bile duct exploration (LCBDE) which reflected the advantage of rigid scopes had risen to be a very promising minimally invasive alternative for the treatment of common bile duct (CBD) stone. Currently, there are mainly two kinds of minimally invasive treatments for choledocholithiasis, which refers to the "one-stage" laparoscopic method, LCBDE and the "sequential two-stage" method, ERCP followed by LC. Both methods are able to achieve the same therapeutic purpose. However, there has always been a controversy about the advantages and disadvantages due to lack of evidence from long-term follow-ups, especially the difference of long-term complications related to Oddi's sphincter functional status, which importantly refers to stone recurrence rates and cholangitis.

The potential long-term complications resulted from EST remains an issue now. It is believed that EST handles Oddi's sphincter stenosis, regurgitation cholangitis, and higher cholangiocarcinoma risks in a long run. By virtue of ERCP, multiple high stone clearance rates (87%~97%) were reported, but meanwhile high re-ERCP rates (around 25%) were also indicated because of stone residual, and whether great stone residual rates was linked to future stone recurrence and repeated cholangitis is not clear. Several randomized controlled trial (RCT) studies had compared ERCP plus LC and LCBDE, the results were similar to the aspects of stone removal rates, costs, and patient acceptance. However, the postoperative cholangitis rate of one single center study is quite different from another. Moreover, few studies have related the stone recurrence rate in the long term follow-up. Obviously, previous RCT studies were limited by few comparison of ERCP followed by LC versus LCBDE in long-term complications, especially stone recurrence and cholangitis. Therefore, this multicenter randomize control study is designed prospectively to compare the stone recurrence and cholangitis rates between ERCP plus LC and LCBDE which can reflects the valuable of Oddi's sphincter protection during the disease management, further dedicating the treatment of gallbladder and common duct stone.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years old
* Choledocholithiasis patient did not perform any operation
* Common bile duct stone less than 2cm in maximum diameter

Exclusion Criteria:

* Unwillingness or inability to consent for the study
* Coagulation dysfunction (INR> 1.3) and low peripheral blood platelet count (<50×109 / L) or using anti-coagulation drugs
* Previous EST, EPBD or percutaneous transhepatic biliary drainage (PTBD)
* Prior surgery of Bismuth Ⅱ and Roux-en-Y
* Benign or malignant CBD stricture
* Preoperative coexistent diseases: acute pancreatitis, GI tract hemorrhage, severe liver disease, primary sclerosing cholangitis (PSC), septic shock
* Combined with Mirizzi syndrome and intrahepatic bile duct stones
* Malignancies
* Biliary-duodenal fistula confirmed during ERCP
* Pregnant women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Common bile duct stone recurrence | Up to 5 years
  Stone was diagnosed by MRI or CT whenever be confirmed after 3 months after procedures.

SECONDARY OUTCOMES:
The proportion of patients with all stones removed | Up to 8 hours
Operation time | Up to 8 hours
  For arm1 (LCBED): the whole process of the operation; for arm2 (LC+ERCP): the total of the two procedures, LC and ERCP
Length of stay in hospital | Up to 60 days
The total hospitalization costs | Up to 60 days
Upper abdominal pain after each procedure by Numerical Rating Scale | Up to 60 days
Hemorrhage | Up to 60 days
  Maintained positive fecal occult blood test appears or Hb decreased by 10g/l
Perforation | Up to 7 days
  CT scan shows retroperitoneal space fluid or gas
Acute cholangitis | Up to 5 years
  Intermittent chills and fever after procedures
Bile leakage | Up to 60 days
  Any bile juice aspirated from the abdominal cavity after procedures
Stricture of the bile duct | Up to 5 years
  Any stricture appears after the procedures
Number of Death connected with the procedures and complications | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Xun Li, M.D., Ph.D., Principal Investigator — Hepatopancreatobiliary Surgery Institute of Gansu Province
Locations (12):
- China (12):
  - The first hospital of Lanzhou University, Lanzhou, Gansu
  - Union hospital,Tongji medical collage,Huazhong University of science and technology, Wuhan, Hubei
  - Second Xiangya Hospital, Central South University, Changsha, Hunan
  - The First Hospital of Jilin University, Changchun, Jilin
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Shandong jiaotong Hospital, Jinan, Shandong
  - The first affiliated hospital of Xi 'an jiaotong university, Xi’an, Shanxi
  - The First Teaching Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The First Affiliated Hospital, Zhejiang University, Hangzhou, Zhejiang
  - Southwest Hospital of Third Military Medical University, Chongqing
  - Xin Hua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai
  - Tianjin Nankai Hospital, Tianjin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cuschieri A, Lezoche E, Morino M, Croce E, Lacy A, Toouli J, Faggioni A, Ribeiro VM, Jakimowicz J, Visa J, Hanna GB. E.A.E.S. multicenter prospective randomized trial comparing two-stage vs single-stage management of patients with gallstone disease and ductal calculi. Surg Endosc. 1999 Oct;13(10):952-7. doi: 10.1007/s004649901145. PMID 10526025
- [Background] Goh ES, Liang B, Fook-Chong S, Shahidah N, Soon SS, Yap S, Leong B, Gan HN, Foo D, Tham LP, Charles R, Ong ME. Effect of location of out-of-hospital cardiac arrest on survival outcomes. Ann Acad Med Singap. 2013 Sep;42(9):437-44. PMID 24162318
- [Background] Koc B, Karahan S, Adas G, Tutal F, Guven H, Ozsoy A. Comparison of laparoscopic common bile duct exploration and endoscopic retrograde cholangiopancreatography plus laparoscopic cholecystectomy for choledocholithiasis: a prospective randomized study. Am J Surg. 2013 Oct;206(4):457-63. doi: 10.1016/j.amjsurg.2013.02.004. Epub 2013 Jul 17. PMID 23871320
- [Background] Bansal VK, Misra MC, Garg P, Prabhu M. A prospective randomized trial comparing two-stage versus single-stage management of patients with gallstone disease and common bile duct stones. Surg Endosc. 2010 Aug;24(8):1986-9. doi: 10.1007/s00464-010-0891-7. Epub 2010 Feb 5. PMID 20135172
- [Background] Jeon TY, Han ME, Lee YW, Lee YS, Kim GH, Song GA, Hur GY, Kim JY, Kim HJ, Yoon S, Baek SY, Kim BS, Kim JB, Oh SO. Overexpression of stathmin1 in the diffuse type of gastric cancer and its roles in proliferation and migration of gastric cancer cells. Br J Cancer. 2010 Feb 16;102(4):710-8. doi: 10.1038/sj.bjc.6605537. Epub 2010 Jan 19. PMID 20087351
- [Background] Noble H, Tranter S, Chesworth T, Norton S, Thompson M. A randomized, clinical trial to compare endoscopic sphincterotomy and subsequent laparoscopic cholecystectomy with primary laparoscopic bile duct exploration during cholecystectomy in higher risk patients with choledocholithiasis. J Laparoendosc Adv Surg Tech A. 2009 Dec;19(6):713-20. doi: 10.1089/lap.2008.0428. PMID 19792866
- [Background] Sgourakis G, Karaliotas K. Laparoscopic common bile duct exploration and cholecystectomy versus endoscopic stone extraction and laparoscopic cholecystectomy for choledocholithiasis. A prospective randomized study. Minerva Chir. 2002 Aug;57(4):467-74. PMID 12145577